CLINICAL TRIAL: NCT04243265
Title: Clinical Study Relating to Patients Undergoing Medial Femoral Patellar Ligament Reconstruction (MPFL) With Fascia Lata Allograft: 10-year Follow-up.
Brief Title: Clinical Study Relating to Patients Undergoing Medial Femoral Patellar Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPFL
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Patellofemoral Dislocation
Keywords: Patellofemoral Dislocation; MPFL reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with MPFL reconstruction (Experimental): Patients underwent MPFL reconstruction using a minimally invasive technique using a fascia lata allograft performed at the Rizzoli Orthopedic Institute between 2011 and 2015 by the team of Prof. Marcacci.
  Clinical and radiographic evaluation will be performed during outpatients visits.
  Interventions: Procedure: MPFL reconstruction with fascia lata allograft

INTERVENTIONS:
Procedure: MPFL reconstruction with fascia lata allograft — Reconstruction of MPFL using a fascia lata allograft. The rationale for this technique is to stabilize the patella and limit medium to long-term patellofemoral arthritic degeneration by restoring the MPFL in the most anatomical way possible, not using a tubular graft but an aponeurosis with biomechanical characteristics similar to the native MPFL. The MPFL reconstruction can be used alone or in association with the realignment of the extensor apparatus by transposition of the anterior tibial tuberosity, managing to correct most of the recurrent patellofemoral instabilities. Only in very serious particular cases is it necessary to perform more invasive additional procedures with a more uncertain clinical result (such as Trocleoplasty).

SUMMARY:
The objective of the present study will be to evaluate the clinical patellofemoral joint function (primary endpoint) and radiographically the patellofemoral arthritic degeneration (secondary endpoint) of of MPFL reconstruction with fascia lata allograft at a minimum follow-up of 2, 5 and 10 years in a group of 25 patients.

DETAILED DESCRIPTION:
Patellofemoral disorders make up about 20% of all knee pathologies and are often a source of diagnostic and therapeutic doubts for the orthopedic surgeon. In fact, the origin of this type of disorder is multifactorial and they can occur in the form of a large variety of clinical pictures with different penetrance in each patient.

In accordance with the classification of Dejour et al., the instability of the patella can be divided into traumatic and a-traumatic (recurrent or habitual). The latter patients may present a variety of anatomical anomalies that predispose to dislocation: patella hypoplasia, genu recurvatum, conditions of ligament hyperlassity, hypoplastic external femoral condyle, trochlear dysplasia, high patella, torsional defects of the lower limb.

The incidence of patella dislocation is estimated to be 5.8 cases per 100,000 people, with values that become five times higher in patients aged between 10 and 17 years. Conservative treatment is preferable in the first case of acute dislocation, however the recurrence of this episode occurs in a percentage equal to 15 - 44% in these subjects.

Many surgical interventions have been described to correct the various factors that predispose to patellofemoral instability, with variable success rates (72% with the Hauser technique and 93% with the Roux-Goldthwait technique, 73% with that of Fielding et at. and 78% with that of Trillat. after a long follow-up.

On the other hand, Crosby and Insall, Arnbjornsson et al. and Marcacci et al. have demonstrated a similar clinical outcome in long-term controlled studies but an increase in degenerative changes in operated patients compared to patients treated conservatively. This can be explained by the fact that often a single procedure is not sufficient on its own to resolve such a complex pathology, or with the fact that the operations used so far excessively increase the pressures on the patellofemoral cartilage with subsequent arthrosic degeneration.

The medial patello-femoral ligament (MPFL) is one of the main stabilizers of the patella in its movement on the femur; numerous studies have recently shown that this ligament is damaged in almost all cases, thus recognizing the role of structure that most limits the patella in its lateral dislocation to the MPFL (biomechanically speaking about 50 - 60% of the force). Following these studies, the reconstruction of the MPFL as an elective treatment for relapsing patella dislocation has recently been proposed. Currently, countless surgical techniques have been proposed that use various types of grafts: autologous tendons (the first in 1990 from Suganuma et al.), donor tendons (allograft) and synthetic ligaments.

Our team recently developed a minimally invasive MPFL reconstruction technique using an allograft tendon of the fascia lata. The rationale for this technique is to stabilize the patella and limit medium-long term patellofemoral arthritic degeneration by restoring the MPFL in the most anatomical way possible, not using a tubular graft but an aponevrosis with biomechanical characteristics similar to the MPFL native. The MPFL reconstruction can be used alone or in association with the realignment of the extensor system by transposition of the anterior tibial tuberosity, managing to correct most of the recurrent patellofemoral instabilities. Only in very serious particular cases is it necessary perform additional procedures that are more invasive and have a more uncertain clinical result (such as Trocleoplasty).

The objective of the present study will be to evaluate the clinical patellofemoral joint function (primary endpoint) and radiographically the patellofemoral arthritic degeneration (secondary endpoint) of of MPFL reconstruction with fascia lata allograft at a minimum follow-up of 2, 5 and 10 years in a group of 25 patients.

Sample is represented by 25 patients underwent MPFL reconstruction using a minimally invasive technique using a donor-sided fascia tendon (allograft) performed at the Rizzoli Orthopedic Institute between 2011 and 2015 by the team of Prof. Marcacci.

Any concomitant treatments: treatment of associated meniscal lesions (meniscectomy), reconstruction of the anterior cruciate ligament (ACL), realignment of the extensor system by transposition of the anterior tibial tuberosity (intervention by Elmsile-Trillat).

Follow-up visit will be carried out at 2, 5 and 10 years of average follow-up. The "non parametric Wilcoxon" and "paired Student's t-test" tests will be used to determine the changes between the various follow-up intervals in the outcome measurements respectively for the non-parametric variables (Tegner activity level) and for the parametric ones ( SF-12 test, VAS pain test, KOOS test, Kujala test, "tilt" and "sulcus" angles, "Insall-Salvati" report).

The changes between the various follow-up intervals in the objective IKDC score and in the Iwano score will be assessed by means of the "Pearson chi-square test".

All "p values" will be 2-tailed; the significance level will be defined at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* The potential person is of legal age, capable of providing informed consent and must sign the Informed Consent Form approved by the Ethics Committee (EC).
* Diagnosis of MPFL injury, performed before surgery, documented by Magnetic Resonance Imaging (MRI) of the affected knee.
* Absence of osteochondral lesions larger than 3 cm2 at the baseline.
* The contralateral knee was and is asymptomatic, stable and functional.
* The patient must be physically and mentally inclined and must have completed post-operative rehabilitation according to the protocol provided at the time of discharge.

Exclusion Criteria:

* Local or systemic infection
* Knee osteoarthritis documented radiographically at baseline
* Articular cartilage injury greater than grade I of Outerbridge detected during surgery.
* History of anaphylactic reaction.
* Systemic therapy with all types of corticosteroids or immunosuppressants in the 30 days prior to surgery.
* Evidence of osteonecrosis in the involved knee.
* History of rheumatoid arthritis, inflammatory arthritis or autoimmune pathologies.
* Neurological pathologies or conditions that the patient is unsuitable for the rehabilitation protocol.
* Untreated meniscal tissue loss greater than 50% at baseline.
* State of pregnancy.
* Obese or with body mass index BMI> 30 kg / m2.
* Association of Trocleoplasty (intervention that produces degenerative changes in the joint in high apercent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 120 months
  It is a straight line with one end (score 0) meaning no pain and the other end (score 10) meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels.
Short-Form 12 | 120 months
  The SF-12 (Short form health survey) is a questionnaire that aims to investigate the perception of individuals' psychophysical conditions. It is taken from a larger version, the SF-36. It is designed to have similar performance to the SF-36, while taking less time to complete.
  Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
Kujala knee Score | 120 months
  The Kujala score is a 13-item questionnaire for the patient-reported assessment of anterior knee pain. Score interval is between 0 (worse result) 100 points (better result)
Level of Tegner activity | 120 months
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer
Objective evaluation of the International Knee Documentation Committee | 120 months
  The International Knee Documentation Committee (IKDC Questionnaire) is a knee-specific patient-reported outcome which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). It's considered to be one of the most reliable outcome reporting tools in its category and was one of the instruments used in the popular MOON study. IKDC has been subjected to rigorous statistical evaluation and has proven to be a valid and responsive patient-reported outcome measure (PROM).
  Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).

SECONDARY OUTCOMES:
Degree of patello-femoral arthritic degeneration | 120 months
  The radiographic evaluation involves the execution of 3 radiographic projections of the operated knee (lateral projection, axial projection of patella at 30° of knee flexion and long-leg standing radiographs.
  Radiographs will be evaluated by one independent expert radiologist to determine the degree of patello-femoral arthritic degeneration according to the Iwano radiographic scale.
  Stage 0 is normal; stage 1 is mild, in which the joint space is at least 3 mm; stage 2 is moderate, in which the joint space is less than 3 mm, but there is no bony contact; stage 3 is severe, in which partial bony contact less than one-quarter of the joint surface is present; and stage 4 is very severe, in which the joint bony surfaces entirely touch each other.
Patellar tilt angle | 120 months
  The tilt angle is defined as the angle subtended by a line joining the medial and lateral edges of the patella and the horizontal, measured on axial projection of patella at 30° of knee flexion.
Sulcus angle | 120 months
  Angle formed between lines joining the highest points of the bony medial and lateral condyles and the lowest bony point of the intercondylar sulcus, measured on axial projection of patella at 30° of knee flexion.
Insall Salvati ratio | 120 months
  The Insall-Salvati ratio or index is the ratio of the patella tendon length respect to the length of the patella.
  This can be measured on a lateral knee x-ray, with the knee 30 degrees flexed.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Zaffagnini, MD, PhD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crosby EB, Insall J. Recurrent dislocation of the patella. Relation of treatment to osteoarthritis. J Bone Joint Surg Am. 1976 Jan;58(1):9-13. PMID 1249117
- [Result] Arnbjornsson A, Egund N, Rydling O, Stockerup R, Ryd L. The natural history of recurrent dislocation of the patella. Long-term results of conservative and operative treatment. J Bone Joint Surg Br. 1992 Jan;74(1):140-2. doi: 10.1302/0301-620X.74B1.1732244.
- [Result] Chrisman OD, Snook GA, Wilson TC. A long-term prospective study of the Hauser and Roux-Goldthwait procedures for recurrent patellar dislocation. Clin Orthop Relat Res. 1979 Oct;(144):27-30. PMID 535237
- [Result] Dejour H, Walch G, Neyret P, Adeleine P. [Dysplasia of the femoral trochlea]. Rev Chir Orthop Reparatrice Appar Mot. 1990;76(1):45-54. French. PMID 2140459
- [Result] Desio SM, Burks RT, Bachus KN. Soft tissue restraints to lateral patellar translation in the human knee. Am J Sports Med. 1998 Jan-Feb;26(1):59-65. doi: 10.1177/03635465980260012701. PMID 9474403
- [Result] Fielding JW, Liebler WA, Krishne Urs ND, Wilson SA, Puglisi AS. Tibial tubercle transfer: a long-range follow-up study. Clin Orthop Relat Res. 1979 Oct;(144):43-4. PMID 535248
- [Result] Hautamaa PV, Fithian DC, Kaufman KR, Daniel DM, Pohlmeyer AM. Medial soft tissue restraints in lateral patellar instability and repair. Clin Orthop Relat Res. 1998 Apr;(349):174-82. doi: 10.1097/00003086-199804000-00021. PMID 9584380
- [Result] Hefti F, Muller W, Jakob RP, Staubli HU. Evaluation of knee ligament injuries with the IKDC form. Knee Surg Sports Traumatol Arthrosc. 1993;1(3-4):226-34. doi: 10.1007/BF01560215. PMID 8536037
- [Result] Iwano T, Kurosawa H, Tokuyama H, Hoshikawa Y. Roentgenographic and clinical findings of patellofemoral osteoarthrosis. With special reference to its relationship to femorotibial osteoarthrosis and etiologic factors. Clin Orthop Relat Res. 1990 Mar;(252):190-7. PMID 2302884
- [Result] Kodraliu G, Mosconi P, Groth N, Carmosino G, Perilli A, Gianicolo EA, Rossi C, Apolone G. Subjective health status assessment: evaluation of the Italian version of the SF-12 Health Survey. Results from the MiOS Project. J Epidemiol Biostat. 2001;6(3):305-16. doi: 10.1080/135952201317080715. PMID 11437095
- [Result] Kujala UM, Jaakkola LH, Koskinen SK, Taimela S, Hurme M, Nelimarkka O. Scoring of patellofemoral disorders. Arthroscopy. 1993;9(2):159-63. doi: 10.1016/s0749-8063(05)80366-4. PMID 8461073
- [Result] Marcacci M, Zaffagnini S, Iacono F, Visani A, Petitto A, Neri NP. Results in the treatment of recurrent dislocation of the patella after 30 years' follow-up. Knee Surg Sports Traumatol Arthrosc. 1995;3(3):163-6. doi: 10.1007/BF01565476. PMID 8821272
- [Result] Monticone M, Ferrante S, Salvaderi S, Rocca B, Totti V, Foti C, Roi GS. Development of the Italian version of the knee injury and osteoarthritis outcome score for patients with knee injuries: cross-cultural adaptation, dimensionality, reliability, and validity. Osteoarthritis Cartilage. 2012 Apr;20(4):330-5. doi: 10.1016/j.joca.2012.01.001. Epub 2012 Jan 10. PMID 22285738
- [Result] Outerbridge RE. The etiology of chondromalacia patellae. 1961. Clin Orthop Relat Res. 2001 Aug;(389):5-8. doi: 10.1097/00003086-200108000-00002. No abstract available. PMID 11501822
- [Result] Smith TO, Walker J, Russell N. Outcomes of medial patellofemoral ligament reconstruction for patellar instability: a systematic review. Knee Surg Sports Traumatol Arthrosc. 2007 Nov;15(11):1301-14. doi: 10.1007/s00167-007-0390-0. Epub 2007 Aug 8. PMID 17684729
- [Result] Suganuma J, Mochizuki R, Shibata R, Sugiki T, Kitamura K, Tani H, Hasegawa M. Reconstruction of the Medial Patellofemoral Ligament With Arthroscopic Control of Patellofemoral Congruence Using Electrical Stimulation of the Quadriceps. Arthrosc Tech. 2016 Jun 20;5(3):e649-56. doi: 10.1016/j.eats.2016.02.022. eCollection 2016 Jun. PMID 27656392
- [Result] Tegner Y, Lysholm J. Rating systems in the evaluation of knee ligament injuries. Clin Orthop Relat Res. 1985 Sep;(198):43-9. PMID 4028566
- [Result] TRILLAT A, DEJOUR H, COUETTE A. [DIAGNOSIS AND TREATMENT OF RECURRENT DISLOCATIONS OF THE PATELLA]. Rev Chir Orthop Reparatrice Appar Mot. 1964 Nov-Dec;50:813-24. No abstract available. French. PMID 14256559
- [Result] Zaffagnini S, Colle F, Lopomo N, Sharma B, Bignozzi S, Dejour D, Marcacci M. The influence of medial patellofemoral ligament on patellofemoral joint kinematics and patellar stability. Knee Surg Sports Traumatol Arthrosc. 2013 Sep;21(9):2164-71. doi: 10.1007/s00167-012-2307-9. Epub 2012 Nov 24. PMID 23179455
- [Result] Zaffagnini S, Grassi A, Marcheggiani Muccioli GM, Luetzow WF, Vaccari V, Benzi A, Marcacci M. Medial patellotibial ligament (MPTL) reconstruction for patellar instability. Knee Surg Sports Traumatol Arthrosc. 2014 Oct;22(10):2491-8. doi: 10.1007/s00167-013-2751-1. Epub 2013 Nov 7. PMID 24196574
- [Result] Zaffagnini S, Marcheggiani Muccioli GM, Grassi A, Bonanzinga T, Marcacci M. Minimally invasive medial patellofemoral ligament reconstruction with fascia lata allograft: surgical technique. Knee Surg Sports Traumatol Arthrosc. 2014 Oct;22(10):2426-30. doi: 10.1007/s00167-014-2940-6. Epub 2014 Mar 22. PMID 24658149